CLINICAL TRIAL: NCT00906568
Title: Clinical Presentation and Bronchial Inflammation of Allergic Bronchopulmonary Aspergillosis (ABPA) in Patients With Cystic Fibrosis
Brief Title: Evaluation of Bronchial Inflammation in Allergic Bronchopulmonary Aspergillosis (ABPA)
Acronym: ABPA
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. Stefan Zielen, Children´s Hospital, Department of Allergy, Pulmunology and Cystic Fibrosis, Goethe University, Frankfurt, Germany
Other Study IDs: KGU-32/09
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2010-10

CONDITIONS: Cystic Fibrosis,
Keywords: Cystic fibrosis; Sensitization to Aspergillus; Bronchial allergen challenge; Induced Sputum; Bronchial inflammation; Small airways disease (SAD)
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum: total Ig-E and RAST, sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sensitized vs non-sensitized: CF with and without SAD defined by MEF25 <50%

SUMMARY:
Chronic bronchial inflammation is an important clinical feature in cystic fibrosis. Approximately 10% of patients with cystic fibrosis suffer from Allergic Bronchopulmonary Aspergillosis. In addition airway inflammation in patients with cystic fibrosis (CF) plays a major role in progression of CF lung disease. In patients with mild disease (Vital capacity >75%) airway inflammation is often under diagnosed.

Severity of allergy against Aspergillus fumigatus will be examined using radioallergosorbent test and skin Prick-test. Subsequently, in patients with established sensitization (RAST ≥ 0.35 IU/mL) a specific bronchial provocation with Aspergillus will be performed. In addition, exhaled nitric oxide,carbon monoxide, exhaled air temperature and inflammatory cells in sputum is measured. 24 hours after bronchial allergen provocation, exhaled NO, CO, air temperature, and bronchial responsiveness is determined and a second sputum obtained.

This study is designed to characterize patients with CF and sensitization against Aspergillus fumigatus in an early stage to prevent pulmonary complications of ABPA. In addition sputum cytokine profiles in CF patients with mild and moderate disease may be different in patients without and with involvement of small airway disease (SAD).

DETAILED DESCRIPTION:
Since symptoms of Bronchopulmonary Aspergillosis are often identical to bacterial infections, the diagnosis is difficult to make. The disease presents with wheezing, pulmonary infiltrates, and bronchiectasis. The most important diagnostic parameters are asthmatic symptoms with obstruction, positive prick test, elevated total IgE, specific IgE and IgG to Aspergillus fumigatus, eosinophilia and radiological findings. Aspergillus fumigatus acts as an allergen Ig-E mediated allergy. Pathophysiological it is assumed that there are two different mechanisms of allergic inflammation. First, there is a direct effect of Aspergillus fumigatus proteases in the alveolar and bronchial epithelium with release of proinflammatory cytokines (IL-8, IL6, MCP-1) and consecutive chemotaxis of inflammatory cells. Second a CD4+ Th2 response with release of IL-4, IL-5 and IL-13. Recently published studies suggest that Aspergillus spores cause the TH2-dependent inflammation directly. So-called Chitinases (part of innate immunity) induce massive IL-13 stimulation. Induction of chitinase activity (CHIT1) leads to an increased remodeling of the lung. It is currently unclear, to which extent Aspergillus-triggered bronchial inflammation in patients with CF is relevant.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 4 and 45 years
* well-known Cystic fibrosis
* Lung function: FEV1 (% pred.) ≥ 70%

Exclusion Criteria:

* age < 4 and > 45 years
* lung function: FEV1 (% pred.)< 70%
* other chronic diseases or infections (e.g., HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol, drug and/or drug abuse
* inability to capture the scale and scope of the study
* participation in another study

Ages: 4 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Outpatients of Department of cystic fibrosis, Goethe University, Frankfurt, Germany
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The characterization of patients with CF and sensitization to Aspergillus fumigatus, and analyzing involvement of small airway disease (SAD) | 1 year

SECONDARY OUTCOMES:
Aspergillus-induced inflammation in sputum using new mediators (IL-8, IL-13, TLR2 and TLR4, LBP and Chitinasen) with the quantitative PCR and protein assay analysis. | 1 year
  In addition planned data analyze: CF-patients will be divided according to their involvement of small airway disease (SAD) into 2 groups: Group 1 without SAD with MEF25 > 50%, Group 2 with SAD with MEF25 < 50% and cell counts and pro-inflammatory cytokines (IL-5, IL-6, IL-8, IL-13, IL-17, INF) measured by quantitative RT-PCR and protein assay will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, MD, Principal Investigator — Goethe-University Frankfurt
Locations (1):
- Goethe-University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] de Oliveira E, Giavina-Bianchi P, Fonseca LA, Franca AT, Kalil J. Allergic bronchopulmonary aspergillosis' diagnosis remains a challenge. Respir Med. 2007 Nov;101(11):2352-7. doi: 10.1016/j.rmed.2007.06.018. Epub 2007 Aug 3. PMID 17689062
- [Background] Knutsen AP, Bellone C, Kauffman H. Immunopathogenesis of allergic bronchopulmonary aspergillosis in cystic fibrosis. J Cyst Fibros. 2002 Jun;1(2):76-89. doi: 10.1016/s1569-1993(02)00033-4. PMID 15463812
- [Background] Stevens DA, Moss RB, Kurup VP, Knutsen AP, Greenberger P, Judson MA, Denning DW, Crameri R, Brody AS, Light M, Skov M, Maish W, Mastella G; Participants in the Cystic Fibrosis Foundation Consensus Conference. Allergic bronchopulmonary aspergillosis in cystic fibrosis--state of the art: Cystic Fibrosis Foundation Consensus Conference. Clin Infect Dis. 2003 Oct 1;37 Suppl 3:S225-64. doi: 10.1086/376525. PMID 12975753
- [Background] Almeida MB, Bussamra MH, Rodrigues JC. ABPA diagnosis in cystic fibrosis patients: the clinical utility of IgE specific to recombinant Aspergillus fumigatus allergens. J Pediatr (Rio J). 2006 May-Jun;82(3):215-20. doi: 10.2223/JPED.1479. Epub 2006 May 26. PMID 16738737
- [Background] Skov M, Pressler T, Jensen HE, Hoiby N, Koch C. Specific IgG subclass antibody pattern to Aspergillus fumigatus in patients with cystic fibrosis with allergic bronchopulmonary aspergillosis (ABPA). Thorax. 1999 Jan;54(1):44-50. doi: 10.1136/thx.54.1.44. PMID 10343631
- [Background] D'Amato G. Role of anti-IgE monoclonal antibody (omalizumab) in the treatment of bronchial asthma and allergic respiratory diseases. Eur J Pharmacol. 2006 Mar 8;533(1-3):302-7. doi: 10.1016/j.ejphar.2005.12.045. Epub 2006 Feb 7. PMID 16464445
- [Background] Kauffman HF. Immunopathogenesis of allergic bronchopulmonary aspergillosis and airway remodeling. Front Biosci. 2003 Jan 1;8:e190-6. doi: 10.2741/990. PMID 12456379
- [Background] Mall MA, Harkema JR, Trojanek JB, Treis D, Livraghi A, Schubert S, Zhou Z, Kreda SM, Tilley SL, Hudson EJ, O'Neal WK, Boucher RC. Development of chronic bronchitis and emphysema in beta-epithelial Na+ channel-overexpressing mice. Am J Respir Crit Care Med. 2008 Apr 1;177(7):730-42. doi: 10.1164/rccm.200708-1233OC. Epub 2007 Dec 13. PMID 18079494
- [Background] Reese TA, Liang HE, Tager AM, Luster AD, Van Rooijen N, Voehringer D, Locksley RM. Chitin induces accumulation in tissue of innate immune cells associated with allergy. Nature. 2007 May 3;447(7140):92-6. doi: 10.1038/nature05746. Epub 2007 Apr 22. PMID 17450126
- [Background] Seibold MA, Donnelly S, Solon M, Innes A, Woodruff PG, Boot RG, Burchard EG, Fahy JV. Chitotriosidase is the primary active chitinase in the human lung and is modulated by genotype and smoking habit. J Allergy Clin Immunol. 2008 Nov;122(5):944-950.e3. doi: 10.1016/j.jaci.2008.08.023. Epub 2008 Oct 9. PMID 18845328
- [Background] Zhu Z, Zheng T, Homer RJ, Kim YK, Chen NY, Cohn L, Hamid Q, Elias JA. Acidic mammalian chitinase in asthmatic Th2 inflammation and IL-13 pathway activation. Science. 2004 Jun 11;304(5677):1678-82. doi: 10.1126/science.1095336. PMID 15192232